CLINICAL TRIAL: NCT00651950
Title: A Flow Monitor for Pediatric Hydrocephalic Shunts - Bench Study of Sensor Alignment Accuracy and Repeatability
Brief Title: Bench Study of Transcutaneous Hydrocephalic Shunt Flow Sensor Alignment Accuracy and Repeatability
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn due to lack of enrollment.
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-HYDRO-1C-H; 2R44NS049680-02 (NIH)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; shunt dysfunction; shunt flow
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Operator Dependence

SUMMARY:
The study hypothesis is that nurses and doctors can use a transcutaneously powered ultrasonic flow sensor to make repeatable and accurate hydrocephalic shunt flow measurements.

The study participants will align the flowmeter probe with a flow sensor hidden under a thick saline pad that simulates skin. A hidden pump will provide a known flow through the flow sensor as the participants make their measurements. Each participant will repeat these measurements over a period of weeks, and the data will tell whether operator skill influences flow measurement accuracy.

DETAILED DESCRIPTION:
The study hypothesis is that a transcutaneously powered ultrasonic flow sensor for hydrocephalic shunts can be repeatedly and accurately read by medical personnel ranging from nurses to senior neurosurgeons.

The test will involve a prototype implantable hydrocephalic shunt flow sensor and readout electronics. The readout electronics use a pickup coil to transcutaneously operate the sensor once the coil is aligned with sensor's inductive coupling coils.

During the test, the shunt flow sensor will be hidden under a thick saline gel pad whose thickness approximates the skin thickness of an older pediatric patient. A syringe pump will provide a known flow rate through tubing connected to the sensor, but the study participants will not know the pump flow setting.

Three neurosurgeons and six floor nurses will perform this study. Each will use the Transonic flowmeter readout to align the pickup coils of the flowmeter with the hidden sensor to make flow measurements.

Each participant will repeat this measurement multiple times over non-consecutive days.

The recorded data will quantify measurement accuracy and repeatability between different operators, and will determine whether operator skill influences flow measurement accuracy.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgeon
* nurse

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three neurosurgeons and six nurses
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Standard deviation of error between operator-measured flow measurements and actual flow measurements. | Daily and weekly

SECONDARY OUTCOMES:
Flow measurement accuracy vs. the number of times the measurement is conducted. | Daily, weekly

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J Drost, BS, MS, Principal Investigator — Transonic Systems Inc.; Bruce A Kaufman, MD, Study Director — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States